CLINICAL TRIAL: NCT05444998
Title: A Prospective, Open-label, Single-arm Phase II Study of Neoadjuvant Ertuzumab Combined With Pyrrolidone and Nab-paclitaxel in Patients With HER2-positive Early and Locally Advanced Breast Cancer
Brief Title: Neoadjuvant Inituomab, Pyrrolidone and Nab-paclitaxel for HER2+Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20222062-C-1
Record Dates: First submitted 2022-06-26; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Pyrrolidinones; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intuzumab + pyrrolidone + nab-paclitaxel (Experimental): Pyrrolidone 400 mg, qd; nab-paclitaxel 125 mg/m2, qw, D1/8/15; inituzumab 6 mg/kg (first dose 8 mg/kg) q3w, D1; 4 cycles in total (q3w as 1 cycle).
  postoperative adjuvant therapy:4 cycles of epirubicin + cyclophosphamide + physician's choice of anti-HER2 targeted therapy.
  Interventions: Drug: Intuzumab, pyrrolidone, nab-paclitaxel

INTERVENTIONS:
Drug: Intuzumab, pyrrolidone, nab-paclitaxel — Pyrrolidone 400 mg, qd; nab-paclitaxel 125 mg/m2, qw, D1/8/15; inituzumab 6 mg/kg (first dose 8 mg/kg) q3w, D1; 4 cycles in total (q3w as 1 cycle).
  The patient's postoperative adjuvant therapy was 4 cycles of epirubicin + cyclophosphamide + physician's choice of anti-HER2 targeted therapy.
  Multiple drug interruptions for adverse events were allowed throughout.

SUMMARY:
explore the efficacy and safety of the combination of nintedanib and paclitaxel in the neoadjuvant treatment of HER2 positive early or locally advanced breast cancer

DETAILED DESCRIPTION:
This study is a prospective, open-label, single-arm clinical study, and it is planned to include 20 treatment-naive patients with HER2-positive early or locally advanced breast cancer (clinical stage IIA ~ IIIC). Neoadjuvant treatment regimen was nituximab + pyrrolidine + nab-paclitaxel. To explore the efficacy and safety of the combination of nintedanib and paclitaxel in the neoadjuvant treatment of HER2 positive early or locally advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. female treatment-naive patients aged ≥ 18 years and ≤ 75 years;
2. ECOG score 0 ~ 1;
3. HER2-positive breast cancer confirmed by pathological examination, defined as an immunohistochemical (IHC) score of 3 + in > 10% of immunoreactive cells or HER2 gene amplification by in situ hybridization (ISH) results (HER2 gene signal to centromere 17 signal ratio ≥ 2.0 or HER2 gene copy number ≥ 6).
4. known hormone receptor status (ER and PgR);
5. The functional level of major organs must meet the following requirements (no blood transfusion, no leukocyte-elevating and platelet-elevating drugs are used 2 before screening):

1) Blood routine neutrophil (ANC) ≥ 1.5 × 109/L; platelet count (PLT) ≥ 90 × 109/L; hemoglobin (Hb) ≥ 90 g/L; 2) Blood biochemical total bilirubin (TBIL) ≤ upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN; alkaline phosphatase ≤ 2.5 × ULN; blood urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 × ULN; 3) echocardiography score (LVEF) ≥ 55%; 4) 12 ECG Fridericia-corrected QT interval (QTcF) < 470 msec; 6. For premenopausal or non-surgically sterile female patients: agree to abstain from sexual intercourse or use effective contraceptive methods during treatment and for at least 7 months after the last dose of the study treatment.

7. Voluntarily join this study, sign the informed consent form, have good compliance and are willing to cooperate with the follow-up.

Exclusion Criteria:

1. stage IV (metastatic) breast cancer;
2. inflammatory breast cancer;
3. Previous anti-tumor therapy or radiotherapy for any malignant tumor, excluding cured cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma and other malignant tumors;
4. concurrent anti-tumor therapy in other clinical trials, including endocrine therapy, bisphosphonate therapy or immunotherapy;
5. Patients who have undergone major surgical procedures unrelated to breast cancer before enrollment, or have not fully recovered from such surgical procedures;
6. severe heart disease or discomfort
7. inability to swallow, intestinal obstruction, or other factors affecting drug administration and absorption;
8. known to have a history of allergy to the drug components of this protocol: a history of immunodeficiency, including HIV test positive, or suffering from other acquired, congenital immunodeficiency diseases, or a history of organ transplantation; 9. pregnant and lactating female patients, female patients with fertility and positive baseline pregnancy test, or patients of childbearing age who are unwilling to take effective contraceptive measures throughout the trial and within 7 months after the study;

10. suffering from serious concomitant diseases or other diseases that will interfere with the planned treatment of concomitant diseases, or any other conditions that the investigator believes that the patient is not suitable for this study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | At the end of Cycle 1 (each cycle is 14 days)
  absence of invasive carcinoma in the breast and axillary lymph nodes, while residual ductal carcinoma in situ was accepted (ypT0orTisypN0)

SECONDARY OUTCOMES:
adverse effects | during the period of neadjuvant chemotherapy,an average of 4 weeks
  Serious adverse effect occur within neoadjuvant chemotherapy

IPD SHARING:
Plan to Share IPD: No